CLINICAL TRIAL: NCT06162845
Title: Smart Soulitions: A Single-blind Randomized Controlled Trial Comparing Smartphone-based Home Exercise to the Paper-based Standard of Care on Pelvic Floor Muscle Weakness Outcomes and Home Exercise Adherence.
Brief Title: Single-blind RCT Comparing Smartphone vs. Paper-based HEP in Pelvic Floor PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Arkansas (Other)
Responsible Party: Principal Investigator, Sarah Walker, Graduate Student enrolled in PhD in Physical Therapy program, University of Central Arkansas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCentralArkansas
Record Dates: First submitted 2023-11-09; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Pelvic Floor Muscle Weakness
Keywords: Smartphone Applications; Home exercise program; Adherence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded to their group allocation and were not aware that another treatment existed until debriefing and unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm recieving free smartohone-based pelvic floor muscle exercise application (Experimental): Smartphone-based home exercise program for performing pelvic floor muscle exercises
  Interventions: Behavioral: A smartphone based application free to download from the google play and iphone store to provide auditory and visual cues and counting for number of perscribed pelvic floor muscle contractions
- Control arm recieving paper-based home exercise program (Active Comparator): Paper-based home exercise program for performing pelvic floor muscle exercises.
  Interventions: Behavioral: Paper-based home exercise program for pelvic floor muscle exercise

INTERVENTIONS:
Behavioral: A smartphone based application free to download from the google play and iphone store to provide auditory and visual cues and counting for number of perscribed pelvic floor muscle contractions — Use of a smartphone-based home exercise application for pelvic floor muscle exercises with visual and auditory feedback for 10 repetitions of pelvic floor contraction endurance holds and 10 repetitions of pelvic floor quick contractions performed three times per day.
  Arms: Experimental arm recieving free smartohone-based pelvic floor muscle exercise application
Behavioral: Paper-based home exercise program for pelvic floor muscle exercise — Written instructions on a piece of paper for 10 repetitions of pelvic floor contraction endurance holds and 10 repetitions of pelvic floor quick contractions performed three times per day.
  Arms: Control arm recieving paper-based home exercise program

SUMMARY:
The goal of this randomized clinical trial is to investigate the impact of a smartphone-based application on patient-reported outcomes for patients with pelvic floor muscle weakness, and the relationship of patient adherence to outcomes in pelvic floor physical therapy compared to the paper-based standard of care.

An additional aim is the exploration and development of two patient-reported questionnaires to enhance understanding of exercise adherence in outpatient pelvic floor physical therapy and smartphone application self-efficacy. These goals will serve to improve practice recommendations for home exercise prescriptions in this patient population.

Participants will be asked to complete 6 patient-reported outcome measures after they complete four, 60-minute long physical therapy treatment sessions conducted one time per week according to the current standard of care for pelvic floor physical therapy.

The experimental group will be given a free pelvic floor muscle exercise application while the control group will be provided with the paper-based standard of care for their home exercise program.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old

  * Referred to outpatient pelvic floor physical therapy for treatment of pelvic floor weakness
  * Generation 5 or later iPhone, Android, or Smart Device
  * Must be willing to receive Push Notification reminders from the application
  * Must have free space on device to download and install app
  * Must have access to the Google Play store or to iOS Apple App Store

Exclusion Criteria:

* ● Not Meeting Inclusion Criteria

  * Pelvic Organ Prolapse Surgery with complications
  * Neurodegenerative Disease
  * History of TBI or CVA with resulting impairment in long- or short-term memory
  * Denervation injury to the pelvic floor
  * Spinal cord injury
  * Pelvic Pain Condition
  * Incapable of Completing Outcomes Questionnaire without caregiver support
  * Unable to speak and read English
  * Current Pregnancy
  * Less than 6 weeks postpartum
  * Researcher judgement

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned female at birth
Enrollment: 33 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory short-form 20 (PFDI-20) | From date of randomization through study completion, an average of 3 months.
  Patient-reported health-related quality of life outcome measures that are widely used for assessment of pelvic floor dysfunction. The minimum score is 0, and the maximum score is 300. HIgher scores indicate higher levels of dysfunction and mean a worse outcome, lower levels indicate less dysfunction and a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Walker, DPT, Principal Investigator — University of Central Arkansas
Locations (1):
- Advanced Physical Therapy, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in pelvic floor muscle weakness, home exercise adherence, and smartphone application use for home exercise adherence. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact Sarah Walker at sarahmwalker86@gmail.com